CLINICAL TRIAL: NCT01243502
Title: A Multiple Dose, Placebo Controlled Study to Assess the Pharmacokinetics, Safety and Tolerability of Topically Administered CT327 in Healthy Male Volunteers
Brief Title: A Study to Assess the Pharmacokinetics, Safety and Tolerability of CT327 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Creabilis SA (Industry)
Collaborators: LCG Bioscience (Unknown)
Responsible Party: Creabilis Therapeutics, Creabilis Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2114/06-CT327
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Safety
MeSH Terms: interventions — pegcantratinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.01% CT327 (or placebo) (Experimental): Six (of eight) subjects received a single topical dose of 0.01% CT327 followed by a 7 day wash-out period. The subjects then received a single topical dose of CT327 on five consecutive days. Two subjects received placebo.
  Interventions: Drug: 0.01% CT327 (or placebo)
- 0.001% CT327 (or placebo) (Experimental): Six (of eight) subjects received a single topical dose of 0.001% CT327 followed by a 7 day wash-out period. The subjects then received a single topical dose of CT327 on five consecutive days. Two subjects received placebo.
  Interventions: Drug: 0.001% CT327 (or placebo)

INTERVENTIONS:
Drug: 0.01% CT327 (or placebo) — Cream (10 g) was applied at an even thickness over a test area on the back of 10 x 10 cm to give an exposure of 1000 μg/dm2.
  Arms: 0.01% CT327 (or placebo)
Drug: 0.001% CT327 (or placebo) — Cream (10 g) was applied at an even thickness over a test area on the back of 10 x 10 cm to give an exposure of 100 μg/dm2.
  Arms: 0.001% CT327 (or placebo)

SUMMARY:
K-252a is a potent inhibitor of nerve growth factor (NGF) and therefore has the ability to inhibit keratinocyte proliferation. K-252a is strongly lipophilic and therefore passes freely into the cell membranes of keratinocytes and accumulates at a systemic level. In order to reduce the dermal absorption and reduce the possible long-term systemic toxicity this study will assess a PEGylated derivative of K-252a named CT327. This approach should improve the safety profile of the K-252a molecule while maintaining its activity. The primary objective is to assess the safety and tolerability of single and repeat doses of CT327 when applied topically to the skin of healthy male volunteers.

The secondary objective is to evaluate the eventual systemic absorption (pharmacokinetics; PK) of CT327 following single and repeat doses in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject is free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory and other tests.
* The subject is a Caucasian male (Caucasian is defined as having origins in the original peoples of Europe, the Middle East, Western Russia, Afghanistan, or the white racial groups of Africa).
* The subject has a body mass index within the range 19 - 30 kg/m2 and has a weight of ≥ 50 kg.
* The subject is capable of giving informed consent and complying with the restrictions and requirements of the protocol.
* The subject is available to complete the study.
* The subject has been registered with a UK General Practitioner (GP) for 3 months prior to the screening visit.
* A signed and dated consent form has been obtained from the subject in accordance with International Conference on Harmonisation Good Clinical Practice (ICH GCP).

Exclusion Criteria:

* As a result of the medical screening process, the PI or medical delegate considers the subject unfit for the study.
* The subject has significant scars, cuts, wounds, dermal abnormalities, tattoos or naevi in the test areas.
* The subject has a past history of contact dermatitis, psoriasis or keloid.
* The subject has any clinically significant abnormality, in the opinion of the PI, on 12-lead ECGs (including subjects with baseline QTcB > 430 ms) at screening.
* The subject has a history of drug or other allergy that contraindicates his participation.
* The subject has participated in a study with a new molecular entity within 4 months, or any other drug trial within 3 months of dosing with the investigational medicinal product (IMP) or placebo.
* The subject has donated a unit of blood (450 mL) in the 3 months prior to dosing or intends to donate in the month after the last scheduled study visit.
* The subject is currently taking a regular course of medication (including vitamins and herbal remedies).
* The subject regularly, or on average, drinks more than 21 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 125 mL of wine or 20 mL of spirits).
* The subject smokes more than five cigarettes (on average) per day, or has been a smoker of more than 5 cigarettes (on average) per day within the 3 months prior to screening.
* The subject has tested positive for hepatitis B surface antigen, hepatitis C antibody or HIV 1 and 2 antibodies.
* The subject has a history of drug abuse or has tested positive for drugs of abuse at pre-study screening. The subject has a positive screen for alcohol and / or drugs of abuse on admission prior to the first dose.
* The subject has consumed methylxanthine-containing food or beverages (e.g. coffee, tea, cola, chocolate, "powerdrinks", caffeine-containing cold remedies) in the 72 h prior to drug administration.
* The subject has used any prescription medication within 2 weeks or 5 half-lives (whichever is longer) of dosing.
* The subject has used non-prescription medication (e.g. aspirin, vitamins and herbal and dietary supplements) within 7 days prior to dosing, or 14 days if the medication contains grapefruit / grapefruit juice or St John's Wort.
* The subject (including those who have had a vasectomy) does not agree to use barrier contraception (condoms) when engaging in sexual activity with women of child bearing potential during the study and for 90 days after completion of the study.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety as defined by local tolerability, subject incidence of TEAEs, and clinically significant changes in lab safety tests, ECGs, vital signs and PE findings. | 2 weeks
  Each subject received a single topical dose of CT327 (or placebo) followed by a single topical dose of CT327 (or placebo) on five consecutive days with a washout period of 7 days between the two dosing periods.

SECONDARY OUTCOMES:
Pharmacokinetic | 2 weeks
  The secondary endpoint is determination of eventual CT327 plasma levels. PK blood sampling day 1: 0 h, 2 h, 4 h, 6 h, 12 h, 24 h, and 2 h post dose on days 9, 10, 11, 12 and 13.